CLINICAL TRIAL: NCT04329689
Title: Hypertrophic ObsructiveCardiomyopathy:Should the Mitral Valve be Addressed During Septal Myectomy?
Brief Title: Hyp Obst Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Abdelkareem Hussein, Doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HHosp
Record Dates: First submitted 2020-03-05; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- septal myectomy alone versus septal myectomy (Experimental): The aims of the present study is to:
  1. Compare the results of adequate septal myectomy alone versus septal myectomy + mitral repair in patients with HOCM.
  2. Effect of mitral repair on outcome of patients with systolic anterior motion that accompanies HOCM.
  Interventions: Other: The Septal myectom

INTERVENTIONS:
Other: The Septal myectom — The Septal myectomy is the preferred treatment of most patients with HOCM, and many studies have documented relief of symptoms and satisfactory late patient survival after relief of outflow tract gradients.
  valve repair or replacement may be necessary

SUMMARY:
Hypertrophic Obstructive cardiomyopathy (HOCM) is the most common genetic cardiomyopathy, heterogeneous in phenotype and clinical course. The genotype-phenotype relationship and associated molecular mechanisms are still incompletely understood. In the HOCM milieu, increased energy cost of force production, impairing performance and mitochondrial function, may be associated to patients' genotype and/or phenotype

DETAILED DESCRIPTION:
Hypertrophic Obstructive cardiomyopathy (HOCM) is the most common genetic cardiomyopathy, heterogeneous in phenotype and clinical course. The genotype-phenotype relationship and associated molecular mechanisms are still incompletely understood. In the HOCM milieu, increased energy cost of force production, impairing performance and mitochondrial function, may be associated to patients' genotype and/or phenotype (1).

Hypertrophic cardiomyopathy as a clinical entity was first described by Brock in 1957 (2). Hypertrophic cardiomyopathy is the most common cause of sudden cardiac death in young people, including competitive athletes (3).

The characteristic pathologic features of hypertrophic cardiomyopathy are asymmetric hypertrophy, especially of the interventricular septum myocardial fiber hypertrophy and disorganisation of myocardial cells, abnormal thickened intramyocardial coronary vessels ("small vessel disease") and interstitial fibrosis (4). In the majority of patients (approximately 90%), hypertrophy mainly involves the interventricular septum and anterolateral wall. In a minority of patients myocardial hypertrophy is confined to the apical part of the left ventricle (4).

Myocardial hypertrophy is not the only hallmark of hypertrophic Obsructive cardiomyopathy. Klues et al. have described anatomic alterations in the mitral apparatus which may be present in this disorder: an increase of the mitral valve area, increase in length of the anterior leaflet, abnormal laxity and anterior displacement of the valve (5). Mitral valve (MV) leaflets have an important role in the pathophysiological process of left ventricular (LV) outflow tract obstruction in patients with hypertrophic obstructive cardiomyopathy (HOCM). Systolic anterior motion (SAM) of the mitral apparatus and contact of the leaflets with the hypertrophied septum narrow the LV outflow, leading to dynamic pressure gradients and in many patients, mitral regurgitation (MR) (6).

Currently, surgery is the gold standard treatment for most drug refractory and severely symptomatic patients [New York Heart Association (NYHA) class III or IV] with obstructive HOCM [7].

The Septal myectomy is the preferred treatment of most patients with HOCM, and many studies have documented relief of symptoms and satisfactory late patient survival after relief of outflow tract gradients.

valve repair or replacement may be necessary (7). However, adequate septal myectomy relieves outflow tract gradients, SAM of the MV, and MR in many patients (6). Nevertheless, several reports have described adjunctive techniques of mitral valvuloplasty aimed at eliminating SAM of the MV (8,9).

Guidelines support decisions to select surgery for patients with mitral structural abnormalities. The 2011 American guidelines state: "Additionally, specific abnormalities of the mitral valve and its support apparatus can contribute significantly to the generation of outflow tract obstruction, suggesting the potential value of additional surgical approaches (e.g., plication, valvuloplasty, and papillary muscle relocation) and making myectomy more appropriate than alcohol septal ablation in some patients" (10)

Finally, An appreciation of mitral abnormalities in HCM has accumulated over the past 20 years (11). There has been a natural response by surgeons to this greater understanding of the contribution of mitral pathology to SAM. At myectomy, they have tried to avoid leaving unrepaired pathology by repairing the mitral valve (12).

ELIGIBILITY:
Inclusion Criteria:

1. All patients that present with hypertrophic obstructive cardiomyopathy (HOCM) with mean pressure gradient>50 mm Hg at rest or on provocation
2. HOCM patients with severe mitral regurgitation.
3. HOCM patients with New York Heart Association (NYHA) functional class II to IV despite optimal medical treatment consisting of -blocking agents, calcium channel blockers, or both.

Exclusion Criteria:

b. Exclusion criteria:

1. Non-obstructive physiological characteristics.
2. Previous MV surgery.
3. Patient with intrinsic pathology of the mitral valve.
4. Patients <18 years.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
LVOT obstruction degree in cm by Echocardiography | 3 months
  The degree of the LVOT obstruction as measured in cm by echocardiography .
Systolic anterior motion of mitral valve | 3 months
  The presence of systolic anterior motion of mitral valve as assessed by post-operative echocardiography.

SECONDARY OUTCOMES:
Post-Operative complictions | 3 months
  Post-operative assessment by echocardiography for complications such as mitral regurgitation.
post-operative general condition | 3 Months
  Assessment of post-operative general condition in terms of NYHA Classification.
Post-operative mortality | 3 months
  assessment of post-operative mortality rate